CLINICAL TRIAL: NCT06215001
Title: Individualized Selection of PEEP in Patients Affected by Expiratory Flow Limitation: a Randomized Controlled Trial
Brief Title: Individualized Selection of PEEP in Patients Affected by Expiratory Flow Limitation
Acronym: PEEP-EFL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Savino Spadaro, Principal investigator, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEEP-EFL
Record Dates: First submitted 2023-11-06; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Complications; Mechanical Ventilation Complication
MeSH Terms: conditions — Postoperative Complications | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EFL Positive - intervention (Experimental): Patients with Expiratory flow limitation will undergo a positive end-expiratory pressure trial to assess the level of positive end-expiratory pressure that eliminates the Expiratory Flow limitation. Positive end-expiratory pressure will be therefore set according to this value.
  Interventions: Procedure: Mechanical ventilation setting (Positive end-expiratory pressure) according to Expiratory Flow Limitation
- EFL Positive - control group (Active Comparator): Patients with Expiratory flow limitation will undergo a positive end-expiratory pressure trial to assess the level of positive end-expiratory pressure that eliminates the Expiratory Flow limitation. Positive end-expiratory pressure will be set at a fixed level of 4 cmH2O.
  Interventions: Procedure: Mechanical ventilation setting (Positive end-expiratory pressure) not according to Expiratory Flow Limitation
- EFL negative patients (No Intervention): Patients with negative positive end-expiratory pressure test (no expiratory flow limitation) will be treated according to the current evidence and followed up for 7 days after surgery to evaluate the incidence of pulmonary postoperative complications.

INTERVENTIONS:
Procedure: Mechanical ventilation setting (Positive end-expiratory pressure) according to Expiratory Flow Limitation — Positive End expiratory pressure will be set according to the positive end-expiratory pressure able to revert the expiratory flow limitation.
  Arms: EFL Positive - intervention
Procedure: Mechanical ventilation setting (Positive end-expiratory pressure) not according to Expiratory Flow Limitation — Positive End expiratory pressure will be set not according to the positive end-expiratory pressure able to revert the expiratory flow limitation but to a standard level of 4 cmH2O.
  Arms: EFL Positive - control group

SUMMARY:
The goal of this clinical trial is to compare different mechanical ventilation settings in Patients undergoing laparoscopic surgery and affected by Expiratory flow limitation. The main question[s] it aims to answer are:

* If individualizing mechanical ventilation on expiratory flow limitation can reduce pulmonary postoperative complications;
* If patients with expiratory flow limitation have a higher incidence of pulmonary postoperative complications as compared to patients with no expiratory flow limitation;

Participants will be screened for expiratory fow limitation and patients with positive screening will be randomized into two groups. Each group will receive a different intraoperative mechanical ventilation:

* Personalized positive end-expiratory pressure based on EFL
* Standard of care positive end-expiratory pressure

Researchers will then compare the two groups to see if the incidence of pulmonary postoperative complications in the first 7 days after surgery is different.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 90 years old;
* Patients undergoing laparoscopic, robotic surgery
* Surgery performed in elective regimen;
* Length of mechanical ventilation more than 120 minutes;
* Presence of invasive pressure monitoring for clinical purposes;

Exclusion Criteria:

* Age < 18 or > 90;
* Severe chronic obstructive pulmonary disease with GOLD stage 3 or 4;
* Length of mechanical ventilation less than 120 minutes;
* Unplanned conversion to laparotomy surgery;
* Refusal to participate by the patient;
* Anesthesia maintenance using Desflurane.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1536 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | First 7 days after surgery
  The investigators will evaluate the number of Pulmonary postoperative complications in the first 7 days after surgery

SECONDARY OUTCOMES:
Postoperative Oxygenation | Within 2 hours after surgery
  The investigators will evaluate postoperative oxygenation after surgery
Need for intubation or non-invasive ventilation | First 7 days after surgery
  The investigators will evaluate the need for intubation or non-invasive ventilation
Days of hospitalization | From hospital entrance to hospital discharge, assessed up to 30 days
  The investigators will evaluate the number of days of hospital stay
Need for Intensive Care admission | From hospital entrance to hospital discharge, assessed up to 30 days
  The investigators will evaluate the need for Intensive Care admission
Length of stay in ICU | From intensive care entrance to intensive care discharge, assessed up to 30 days
  The investigators will evaluate the length of Intensive care unit stay

IPD SHARING:
Plan to Share IPD: Undecided